CLINICAL TRIAL: NCT01441310
Title: Laparoscopic Sentinel Node Navigation Surgery for Gastric Cancer
Acronym: SNNS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Ho Kim, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBHGS01
Record Dates: First submitted 2011-09-25; First posted 2011-09-27 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Sentinel node navigation surgery; Dual method; Recurrence
MeSH Terms: conditions — Stomach Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic sentinel node navigation surgery (Experimental): Laparoscopic sentinel node navigation surgery
  Interventions: Procedure: Laparoscopic sentinel node navigation surgery

INTERVENTIONS:
Procedure: Laparoscopic sentinel node navigation surgery — Laparoscopic SNNS using simultaneous indocyanine green (ICG) and 99mTc-antimony sulfur colloid (ASC) injections

SUMMARY:
There are few reports on a dual dye and isotope approach using laparoscopy in gastric cancer sentinel node mapping.

The aim of this study was to evaluate the feasibility of laparoscopic limited gastrectomy with sentinel basin(SB) dissection for gastric cancer using simultaneous indocyanine green (ICG) and 99mTc-antimony sulfur colloid (ASC) injections.

DETAILED DESCRIPTION:
Prospective phase II clinical trials for sentinel node navigation surgery(SNNS) in early gastric cancer.

Laparoscopic SNNS:

1. ICG and 99mTc-antimony sulfur colloid (ASC) submucosal injection under intraoperative endoscopy
2. Sentinel node basin identification and dissection
3. Sentinel nodes picking in back table
4. Frozen biopsy of sentinel nodes(hematoxylin and eosin staining and immunohistochemistry for cytokeratin)
5. If the sentinel node biopsy by frozen section is negative, limited gastrectomy will be performed or if positive, radical D2 gastrectomy will be performed.

Sample size: 100 cases

Study duration: 5 years( 2year enrollment, 3 year follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Age 20-80
* Informed consent
* No other malignancies
* cT1N0 stage gastric cancers < 4cm
* no allergic history of isotope

Exclusion Criteria:

* Patients eligible for endoscopic submucosal dissection(ESD) with absolute indication

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
3 Year disease free survival | Postoperative 3 year
  Recurrence evaluation by eddoscopy, computed tomography and Positron emission tomography if needed.

SECONDARY OUTCOMES:
Sentinel node detection rate, occurrence of complication ,Qualtity of life and remnant stomach function evaluation. | postoperative 1, 3, 6, 12 month
  Sentinel node detection rate and occurrence of complication of SNNS using dual method for gastric cancer were evaluated QoL questennaire and remnant stomach function were evaluated for the evaluation of patient's quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Ho Kim, M.D.Ph.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No